CLINICAL TRIAL: NCT04395391
Title: Usability Study of Home Collection and Mailing With SARS-CoV-2 Test Specimen Collection Materials (2020-06)
Brief Title: Home Usability Study of the SARS-CoV-2 (COVID-19) Test
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-06
Record Dates: First submitted 2020-05-19; First posted 2020-05-20 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
Keywords: COVID-19; Sample Collection; Human Factors Study; Nasal Swab
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples may be retained for purposes such as additional testing in this or alternative SARS-CoV-2 tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 — Determine usability of study materials and kit

SUMMARY:
The primary objective is to determine the usability of the SARS-CoV-2 Specimen Collection Materials for at-home collection and mailing of sample to the testing laboratory.

DETAILED DESCRIPTION:
This study is a prospective observational human factors usability study designed to evaluate the Instructions For Use (IFU) in the SARS-CoV-2 Specimen Collection Materials based on the successful completion of self-collection of a nasal swab sample, which includes a valid SARS-CoV-2 test result.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent

Exclusion Criteria:

* Prior medical or laboratory training
* Prior experience with COVID-19 specimen self-collection
* Prior SARS-CoV-2 testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects of varying education levels, age, and health status. Subjects will be employees of Exact Sciences. Subjects are considered enrolled when they provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-06-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Exact Sciences, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study will be shared after deidentification. This may include text, tables, figures, and appendices. The study protocol, informed consent form (when applicable), and statistical analysis plan (when applicable) will also be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available from 2 years and ending 4 years after publication. Data will be shared with researchers who provide a methodologically sound proposal to achieve the aims outlined in the approved proposal.
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary IRB/EC approvals or waivers as applicable to conduct research. Data will be available between 2 and 4 years after publication through the Sponsor.

RESULTS

PARTICIPANT FLOW:
Groups:
- Volunteers: Men and women who had no prior medical or laboratory training, no prior experience with COVID-19 self-collection, or no prior SARS-CoV-2 testing.
Period: Overall Study
Arm/Group | Volunteers
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Volunteers
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
Level of Education [Count of Participants; unit: Participants]
  College degree, or higher | 23
  Other level of education | 7

OUTCOME MEASURES:

1. Primary Outcome: Valid SARS-CoV-2 Test
Description: The percent of samples from the fully enrolled cohort to return a valid SARS-CoV-2 test result (positive, not detected, or inconclusive)
Time Frame: Subjects are assessed at enrollment
Population: Each participant only completed one test.
Measure: Count of Participants; unit: Participants
Arm/Group | Volunteers
Number analyzed (Participants) | 30
Participants | 30

ADVERSE EVENTS:
Time Frame: Adverse event collection began at enrollment and ended after completion of the sample collection, up to one hour.
Description: Serious adverse events are not expected for this study. All-Cause mortality is not expected for this study.
Arm/Group | Volunteers
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator agreed that they shall not, without the Sponsor's prior written consent, independently publish, publicly disclose, present or discuss any results of or information pertaining to the activities conducted under their agreement for a period of one (1) year following completion of the Study.

DOCUMENTS (3):
  • Study Protocol (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT04395391/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT04395391/SAP_001.pdf
  • Informed Consent Form (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT04395391/ICF_002.pdf